CLINICAL TRIAL: NCT03655782
Title: Retraining Neural Pathways Improves Cognitive Skills After A Mild Traumatic Brain Injury
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Perception Dynamics Institute (Industry)
Collaborators: University of California, San Diego (Other); University of South Alabama (Other); University of California, Riverside (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PerceptionDI
Record Dates: First submitted 2018-08-29; First posted 2018-08-31 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-05

CONDITIONS: MTBI - Mild Traumatic Brain Injury
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Intervention Model Description: The investigators will show that working memory, processing speed, reading speed, and attention improve significantly in mTBI patients after 36 30-minute training sessions of PATH training followed by digit memory exercises for different doses (once, twice or three times a week) to determine which dose improves cognitive skills the most, and whether the improvements are sustained over time. MEG brain imaging will be used to show that PATH neurotraining followed by digit memory exercises improves the function of the dorsal, attention, and working memory networks (e.g., PPC, DLPFC and ACC/PCC areas), reducing over recruitment, as found during Phase I.
Who Masked: Participant, Care Provider
Masking Description: Staff will not be told which treatment group the subject was in.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PATH+DM neurotraining three times a week for 36 30-minute sessions (Experimental): Subject looks at computer screen to determine whether dim gray stripes in fish-shaped window move left or right relative to gray stationary background stripes. The subject reports which way center stripes move by pushing left or right arrow key, receiving brief tone if incorrect. Program adaptively changes the contrast of the test pattern in order to keep subject at 79% correct. There are levels of difficulty introduced by making the background pattern more similar to that in fish, by increasing pattern's complexity level, and by increasing number of directions of movement from one to two directions of motion. Intervention will be trained for 20 minutes, followed by 10 minutes of digit memory exercises 3 times each week for 12 weeks. Ten minutes of digit memory (DM) practice, recalling the correct sequence of digits, each presented for 500 msec, from 5 digits up to 10 digits will be completed for 10 minutes following 20-minutes of PATH neurotraining.
  Interventions: Behavioral: PATH + DigitMemory (DM) neurotraining
- PATH+DM neurotraining two times a week for 36 30-minute sessions (Experimental): Subject looks at computer screen to determine whether dim gray stripes in fish-shaped window move left or right relative to gray stationary background stripes. The subject reports which way center stripes move by pushing left or right arrow key, receiving brief tone if incorrect. Program adaptively changes the contrast of the test pattern in order to keep subject at 79% correct. There are levels of difficulty introduced by making the background pattern more similar to that in fish, by increasing pattern's complexity level, and by increasing number of directions of movement from one to two directions of motion. Intervention will be trained for 20 minutes, followed by 10 minutes of digit memory exercises 2 times each week for 18 weeks. Ten minutes of digit memory (DM) practice, recalling the correct sequence of digits, each presented for 500 msec, from 5 digits up to 10 digits will be completed for 10 minutes following 20-minutes of PATH neurotraining.
  Interventions: Behavioral: PATH + DigitMemory (DM) neurotraining
- PATH+DM neurotraining once a week for 36 30-minute sessions (Experimental): Subject looks at computer screen to determine whether dim gray stripes in fish-shaped window move left or right relative to gray stationary background stripes. The subject reports which way center stripes move by pushing left or right arrow key, receiving brief tone if incorrect. Program adaptively changes the contrast of the test pattern in order to keep subject at 79% correct. There are levels of difficulty introduced by making the background pattern more similar to that in fish, by increasing pattern's complexity level, and by increasing number of directions of movement from one to two directions of motion. Intervention will be trained for 20 minutes, followed by 10 minutes of digit memory exercises once a week for 36 weeks. Ten minutes of digit memory (DM) practice, recalling the correct sequence of digits, each presented for 500 msec, from 5 digits up to 10 digits will be completed for 10 minutes following 20-minutes of PATH neurotraining.
  Interventions: Behavioral: PATH + DigitMemory (DM) neurotraining

INTERVENTIONS:
Behavioral: PATH + DigitMemory (DM) neurotraining — Improve visual timing and sensitivity in the dorsal stream. The mTBI subject will sit 57 cm in front of a computer monitor. During the presentation, the bars in the 'fish-shaped' window in the center of the screen formed by a sinusoidal grating, move left or right very briefly. When the screen goes blank, the subject reports which way the center pattern moved by pushing the left or right arrow key. A brief tone is presented after incorrect responses. The program adaptively changes the contrast of the test pattern so that the subject detects motion at lowest contrast possible. A sequence of patterns in each training cycle that are designed to optimally activate magnocellular neurons are shown to the subject. There are two programs, the first measures the contrast needed to see one direction of movement, and the second program measures the contrast needed to see two directions of movement, requiring memory. Both are followed by digit memory exercises.
  Other Names: PATH to Insight; PATH to Reading

SUMMARY:
The proposed study tests the efficacy (Phase II) of 36 30-minute training sessions of PATH neurotraining followed by digit memory exercises to improve working memory, processing speed and attention in mTBI patients rapidly and effectively to provide clinical testing of a therapeutic training for the remediation of cognitive disorders caused by a concussion. This study will contribute to the fundamental knowledge of how to remediate concussions from a mTBI to enhance the health, lengthen the life and reduce the disabilities that result from a mTBI.

DETAILED DESCRIPTION:
This study will provide clinical testing of therapeutic training for remediation of concussion-induced cognitive disorders. Our Phase I Clinical Trial determined the feasibility of targeting visual timing deficits in mTBI subjects to successfully remediate cognitive deficits. This trial identified PATH+DigitMemory (DM) neurotraining as the most effective intervention for post-mTBI cognitive remediation. Since Institutional Review Boards have classified these cognitive interventions as minimal risk and not yet proven treatments for mTBI, FDA approval is not required before study initiation. Upon protocol approval by Pearl IRB, recruitment materials will be distributed through clinicians with interested TBI patient waitlists. Participants will comprise two mTBI subgroups: 1) those who initially experienced a severe TBI (moderate TBI group) and 2) those with an initial mTBI. Prospective participants will undergo telephone screening to determine study eligibility. Groups will be balanced for age, sex, visual working memory performance, number of TBI incidents, duration of loss of consciousness, and locus/extent of mTBI. We anticipate 3-5 mTBI referrals monthly from community-based sources established during Phase I, facilitating recruitment of 90 mTBI subjects over the three-year study period. This study is designed to enhance understanding of and provide training targeted toward cortical timing processes (PATH+DM training), extending our Phase I findings to a substantially larger mTBI subject sample.

This Phase II research represents a randomized, within-subject clinical trial investigating cognitive and behavioral effects of different training frequencies-36 sessions of 30-minute PATH+DM training (20 minutes PATH followed by 10 minutes Digit Memory exercises) administered once, twice, or three times weekly in adults aged 18-60. We will show that after completing the PATH+DM training, subjects have significantly higher cognitive skills than before. Changes in test performance for the primary outcome variable: VWM, and secondary outcome measures: processing speed, selective attention, cognitive flexibility, AWM, reading speed, and questionnaires will be analyzed using mixed-factors Multivariate Analysis of Variance (MANOVA). These MANOVAS will compare standardized test percentiles, reading rate, and questionnaire scores, controlling for age, before and after PATH+DM neurotraining. The mixed factors MANOVA will be performed with the between-subjects factor of Training Group (PATH+DM training once, twice or three times/week) and the within-subjects factor of Time (Time1, Time2, Time3, and Time4), corresponding to Initial, 3 months, 6 months, and 12 months after starting PATH+DM training, to test the effects of dosage on the magnitude of improvements in cognitive skills (Aim 1). One analysis will be performed for each behavioral test to compare improvements in standardized percentiles, and reading rate scores following PATH+DM on the three different frequencies being investigated. Planned a-priori contrasts are predicted to reveal group differences such that improvements at Time 2 (3 months after starting intervention) will be largest for the PATH group doing PATH 3 times a week. Another question being answered is whether this advantage at Time 2 is also found at Time 3, 6 months after starting intervention. A related question is whether participants who have the lowest scores will also demonstrate the greatest improvements. We expect that those in the moderate TBI group will improve more than those in the mild TBI group for this reason. These answers will help to determine the relative efficacy of PATH training for a wide range of TBI patients who experience memory loss. The results from Aim 1 above, post-tests 3, 6 and 12 months after starting PATH+DM training, will be analyzed with Multi Level Modeling (MLM), a technique particularly well suited for capturing the effects in studies with complex variables that are nested within one another, and that will permit growth curve modeling over multiple measurements. To test whether improvements in cognitive skills after PATH+DM training are sustained over time (Aim 2), we will have measurement periods (x4) nested within the random effect of participants, and the between subjects, fixed effect of conditions of Training Group.

The PATH+DM intervention promotes sustained functional recovery from an mTBI, when currently there are no proven solutions for mTBI: 80% of TBIs. MEG recordings before and after training will provide a biomarker, a neural correlate, to determine whether PATH training improves the function of the dorsal, attention, and working memory networks. Preliminary data suggest that MEG imaging is sensitive in detecting brain functional changes in dlPFC and ACC which are part of the VWM network. MEG may be a unique biomarker of timing deficits in mTBI. MEG pre-post recordings will be examined to understand the distribution of timing-based deficits across a population of mTBI patients. Resting-state MEG is sensitive in detecting neuronal abnormalities in mTBI on an individual-subject basis. We will use MEG functional imaging-based neurophysiological recordings to test whether the dorsal stream visual, attention, and memory networks improve in function significantly more following PATH+DM training than before PATH+DM training (Aim 3). A structural MRI to superimpose the functional activity on top of the brain anatomy will be collected before the initial MEG recording. To evaluate PATH+DM training effectiveness across different doses, we will analyze improvements in MEG neurophysiological recordings during two time intervals: 100-200 milliseconds (examining visual system functional changes) and 200-1000 milliseconds (studying later responses of the working memory network). Voxel-wise MEG neurophysiological recordings will be collected from all qualifying mTBI subjects, serving as a biomarker to demonstrate PATH+DM neurotraining's feasibility for cognitive improvement. Whole-brain MEG images across frequency bands will be analyzed using the Fast-VESTAL procedure to measure time-locked signals during an N-Back working memory task, evaluating brain function improvements as implemented in our pilot studies. We hypothesize that MEG timing deficits will predict which mTBI subjects respond optimally to PATH+DM training, and that subjects demonstrating large MEG recording differences will exhibit the largest behavioral improvements. We further hypothesize that individuals receiving PATH+DM training three times weekly will show significantly stronger neuronal signals, better performance accuracy, and shorter reaction times compared to those training once weekly. We also expect to observe more significant increases in response magnitude and coupled theta/gamma and/or alpha/gamma oscillations following PATH+DM training compared to baseline, as suggested by our pilot studies. These hypotheses will be examined in an expanded participant sample to establish effect sizes for larger cohorts than studied in Phase I, comparing improvement magnitude between moderate and mild TBIs, and assessing whether improvements in different cortical areas persist over time. To increase its commercialization ability, PATH+DM training must be shown to improve brain function using a biomarker, as stated by neurologists and therapists in letters of support.

We will also examine moderators that may determine training outcome (Aim 4). The goal is to use MEG-based neural correlates of timing deficits in conjunction with behavioral cognitive assessments to understand the distribution of timing-based deficits across a population of mTBI subjects, and how these deficits predict cognitive skill deficits, that are moderated by individual factors. We will determine whether individual differences at initial assessment predict improvements following training for different subpopulations: 1) Moderate vs. mild TBI, 2) different age groups (18-28, 29-41, 42-60), 3) concussion frequency, and 4) varying loci and extent of mTBI deficits. We will investigate whether MEG functional imaging-based neurophysiological recordings of timing-based deficits predict cognitive skill deficits, and whether these relationships are moderated by individual factors including concussion frequency, duration of loss of consciousness, nature and extent of cognitive deficits, injury severity (moderate versus mild), and age. Studies incorporating MEG biomarker assessment will establish pre-post timing and functional capabilities of different cortical areas within visual, attention, and executive control pathways, complemented by pre-post behavioral neuropsychological testing of cognitive abilities. This exploratory aim will help determine whether different therapeutic approaches should be developed for different mTBI types and age groups.

Implementation Plan To ensure standardized test administration, written instructions will be delivered verbatim.

Training (PATH+DM) will be conducted using the subject's own computer (Macintosh, Windows, or Chromebook) by the PI either at PDI's Solana Beach office or remotely via Zoom. Training sessions will occur each morning at times convenient for participants to complete 36 training sessions of 30 minutes each, 1-3 days weekly. The PI will implement PATH+DM training with high fidelity, supported by training videos. Each subject will receive one-on-one instruction to ensure proper task execution. The PI will monitor subject engagement by examining computer data and providing additional training when necessary. All sessions will be supervised to ensure consistent implementation at the same time of day. This supervision is essential since mTBI subjects are relearning attention and memory skills, making independent task completion less reliable. Text reminders will be sent to encourage timely attendance. If a subject experiences discomfort (e.g., boredom, mild headache, fatigue, or dizziness) from visual or memory tasks, they will be instructed to look away from the screen and take a brief break. Such side effects are uncommon.

Dr. Lawton, the PI, brings over 45 years of experience conducting controlled validation studies. She will oversee staff training and manage daily operations, including scheduling and supervising pre-post neuropsychological testing and administering PATH+DM training. She will also coordinate MEG examinations at UCSD. To prevent bias, the PI will not be involved in data collection. Staff will collect standardized test data, while the PATH+DM web application will automatically record training data. Behavioral data will be analyzed exclusively by our statistician, Dr. Shelley-Tremblay, who will enter all behavioral test data into REDCap and FITBIR databases and conduct all behavioral data analyses.

Professor Huang and his team will conduct MEG functional imaging-based neurophysiological recordings from all qualifying mTBI subjects to provide biomarker data. Voxel-wise MEG source magnitude images covering the whole brain and each frequency band, following the Fast-VESTAL procedure to measure time-locked signals during an N-back working memory task, will evaluate brain function improvements, replicating methods used in Phase I. These MEG recordings will determine pre-post timing and functional capabilities of different cortical areas in the visual, attention, and executive control pathways, complementing behavioral pre-post standardized neuropsychological assessments of cognitive abilities. A distinctive feature of this study is Dr. Huang's innovative, patented techniques for analyzing MEG functional imaging-based neurophysiological data to detect changes in cognitive function and provide biomarkers for cognitive improvement.

Our team will convene periodically via Zoom to ensure we have a rigorous study implementation and to prepare results for scientific meetings and high-impact journal publications.

ELIGIBILITY:
Inclusion Criteria:

1. Referred by Clinician verifying that patient has an mTBI (also includes moderate TBI: those who had a severe TBI with a loss of consciousness more than 30 minutes that is now an mTBI) and has a visual working memory loss as determined by first neuropsychological pre-test administered: The Test of Information Processing Skills (TIPS),
2. One or more concussions,
3. Any loss of consciousness from 5- 30 min (not longer than 30 min) to be in mTBI group, otherwise in moderate TBI group.
4. Any loss of memory for events immediately before or after the accident for 24 hours is in mTBI group, otherwise is in moderate TBI group,
5. Any alteration of mental state at the time of the accident (e.g. feeling dazed, disoriented, or confused),
6. Be between the ages of 18 to 60 years, when development and aging are not factors,
7. Agrees to complete the study after hearing the time commitment involved,
8. Has corrected 20/20 visual acuity, and normal motor control so can do PATH neurotraining (signal direction that dim gray stripes move by pushing arrow keys on the computer),
9. Can sign and understand the informed consent form themself,
10. Can drive to test sites or capable of using public transportation (bus or train) to test site.
11. Reads English fluently, so can follow instructions.

Exclusion Criteria:

1. mTBI occurred less than 3 months earlier [While post-concussive symptoms (PCS) resolve within days post injury in the majority of individuals with mTBI,127 symptoms can endure 3 months post injury or longer, indicating spontaneous recovery and chronic sequela.128 In the general public, between 8% to 33% of mTBI patients have persistent PCS and long-term cognitive and/or behavioral impairments129 that negatively impact quality of life. In the proposed study, we will try to minimize the confound from the spontaneous recovery by only recruiting chronic mTBI subjects, and not recruiting mTBI subjects with mTBI less than 3 months.] with no maximum time if still experiencing memory problems which will be measured by the TIPS visual working memory (VWM) scores.
2. diagnosis of epilepsy or seizure disorder in last 12 months,
3. diagnosis of moderate depressive disorder or moderate anxiety, having driving limitations in traffic
4. answers 'Yes' to any of the questions on the Columbia Suicide Severity Rating Scale,
5. had a stroke or metabolic derangements causing cognitive impairments, i.e. alcohol or substance abuse,

   And for those chosen to undergo MEG exams:
6. has extensive metal dental hardware (e.g., braces and large metal dentures; fillings are acceptable) or other metal objects in head, neck, or face areas that cause artifacts in MEG data, and are not removable during pre-processing, and
7. has claustrophobia since MRI scanner is in small enclosed space,
8. has a cardiac pacemaker, or 9) is pregnant.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in Visual Working Memory | Immediately before begin intervention and 3, 6, and 12 months later.
  Visual Working Memory (VWM) using Test of Information Processing Skills (TIPS), having two distractor tasks to measure Sequential Processing: the subject must remember a sequence of letters, that are shown one at a time for 2 seconds each, for sequences of from 2 up to 9 letters right after seeing the entire sequence of letters. Short Term that are shown one at a time for 2 seconds each, for sequences of from 2 up to 9 letters right after seeing the entire sequence of letters. Short Term VWM is assessed by recalling the correct sequence of letters after counting from 1 to 10 numbers in sequence, starting at different initial numbers, slowly, and after repeating a short sentence with an animal subject for VWM.
  Delayed Recall is assessed by remembering all animal names in repeated sentences 3 minutes after finish the VWM tests. The TIPS VWM Standardized Percentile Rank goes from <1% to 99%.

SECONDARY OUTCOMES:
Change in Processing Speed | Immediately before begin intervention and 3, 6, and 12 months later.
  Processing Speed using Wechsler Adult Intelligence Scale (WAIS-4) Processing Speed Index (PSI): requires two subtests: 1) the WAIS Symbol Search subtest which requires subjects to scan a target group (two symbols) and search a group of 5 symbols, indicating whether one of the target symbols appears in the search group, and 2) WAIS Digit Symbol Coding subtest, where the subject fills in boxes below digits with symbols that are paired with them in a key at the top of the page. Both of these subtests are timed for two minutes each. The scaled scores from each subtest are combined to create an overall Processing Speed Index score, that is converted to a standardized percentile. WAIS Processing Speed Index Standardized Percentile Rank goes from < 0.1% to > 99%.
Change in Attentional Focus | Immediately before begin intervention and 3, 6, and 12 months later.
  Selective Attention using Delis-Kaplan Executive Function System (DKEFS) Color-Word Interference test measuring time to say color of the printed word that denotes a different color (Stroop test). DKEFS Color-Word Interference Test Standardized Percentile Rank for Inhibition subtest goes from 0.5% to 99.9%.
Change in Cognitive Flexibility | Immediately before begin intervention and 3, 6, and 12 months later.
  Cognitive Flexibility using DKEFS Color-Word Interference test measuring time to switch attention between color of printed word (Stroop test) and printed word when surrounded by a rectangle. DKEFS Color-Word Interference Test standardized scores for Standardized Percentile Rank for Inhibition Switching subtest goes from 0.5% to 99.9%.
Change in Auditory Working Memory | Immediately before begin intervention and 3, 6, and 12 months later.
  Auditory Working Memory (AWM) is assessed using the WAIS-4 Working Memory Index which consists of two subtests: 1) the Digit Span subtest, where the subject has to repeat a list of spoken numbers, requiring the subject to remember subsequently more numbers: in the correct order, backwards, and in numerical sequence on three different subtests, and 2) the Letter-Number Sequencing subtest which requires sequencing subsequently more numbers and letters in the correct numerical and alphabetic sequence. Presentation of the numbers and letters are timed for one second each for these working memory tests. The WAIS Working Memory Index Standardized Percentile Rank goes from < 0.1% to > 99.9%.
Change in Reading Proficiency | Immediately before begin intervention and 3, 6, and 12 months later.
  Using Adult Dyslexia Test, use reading grade level to measure reading proficiency. Evaluates whether a subject's visual processing and phonological processing is markedly, moderately, mildly, or borderline below normal, or is normal or above normal.
Change in DLPFC Function | Immediately before begin intervention and 3, 6, and 12 months later.
  Using the total covariance matrix, voxel-wise MEG source magnitude images that cover the whole brain will be obtained for each subject, and each frequency band, following the Fast-VESTAL procedure, measuring time-locked signals during a working memory N-back task to evaluate improvements in brain function in DLPFC (working memory).
Change in ACC Function | Immediately before begin intervention and 3, 6, and 12 months later.
  Using the total covariance matrix, voxel-wise MEG source magnitude images that cover the whole brain will be obtained for each subject, and each frequency band, following the Fast-VESTAL procedure, measuring time-locked signals during a working memory N-back task to evaluate improvements in brain function in ACC (attention network).
Change in Precuneus/PCC | Immediately before begin intervention and 3, 6, and 12 months later.
  Using the total covariance matrix, voxel-wise MEG source magnitude images that cover the whole brain will be obtained for each subject, and each frequency band, following the Fast-VESTAL procedure, measuring time-locked signals during a working memory N-back task to evaluate improvements in brain function in Precuneus/PCC (attention network).
Change in V1-MT | Immediately before begin intervention and 3, 6, and 12 months later.
  Using the total covariance matrix, voxel-wise MEG source magnitude images that cover the whole brain will be obtained for each subject, and each frequency band, following the Fast-VESTAL procedure, measuring time-locked signals during a working memory N-back task to evaluate improvements in brain function in V1-MT (visual motion network).
Change in Reading Speed | Immediately before begin intervention and 3, 6, and 12 months later.
  Number of words/minute subject can read 6 words of subsequent text from interesting story using computer-based program.
Change in Post-Concussion Symptoms | Immediately before begin intervention and 3, 6, and 12 months later.
  Rivermead Post-Concussion Symptom Questionnaire evaluates 16 symptoms commonly experienced after a concussion, being rated from 0 (not experienced at all) to 4 (a severe problem). The Rivermead PCS evaluates ocular, vestibular, and mental health symptoms of mTBI subject.
Change in Quality of Life | Immediately before begin intervention and 3, 6, and 12 months later.
  ADCS Quality of Life SF-36 questionnaire evaluates subject's general health, activity limitations, emotional health, physical health, social activities, pain, and energy and emotions, having a score from 0-100.
Change in Brain Injury Visual Symptom Survey (BIVSS) | Immediately before begin intervention and 3, 6, and 12 months later.
  BIVSS rates each of 28 visual behaviors by how often each behavior occurs: Never, seldom, occasionally, frequently, or always. The symptoms are in 8 categories: eyesight clarity, visual comfort, doubling, light sensitivity, dry eyes, depth perception, peripheral vision, and reading.

CONTACTS AND LOCATIONS:
Overall Officials: Teri Lawton, Ph.D., Principal Investigator — Perception Dynamics Institute
Locations (2):
- United States (2):
  - University of California at San Diego, San Diego, California
  - Perception Dynamics Institute, Solana Beach, California

IPD SHARING:
Plan to Share IPD: Yes
After completion of the study, deidentified data will be made available to qualified outside investigators following NIH Data Sharing guidelines; none of the data will be considered proprietary. Most of the data for this study will be collected through standardized tests of attention, processing speed, and working memory to be administered by the staff on this project
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: November 2025 for 10 years.
Access Criteria: Qualified investigator